CLINICAL TRIAL: NCT05497479
Title: A Phase 1 Study Evaluating Techniques for Measuring Tear Production
Brief Title: Study Evaluating Techniques for Measuring Tear Production
Acronym: MTP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-110-A
Record Dates: First submitted 2022-07-26; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All eligible subjects will be enrolled and randomized (1:1) to one of two treatment groups: active (0.003% AR-15512) or control (AR-15512 vehicle). Following enrollment, subjects in the two treatment groups will each be randomized 1:1 to which Visit (Visit 1 or 2) anesthetic will be used with the Schirmer test.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with Schirmer test with no anesthetic (Experimental): Both eyes will be treated.
  Interventions: Drug: 0.003% AR-15512 to be administered in both eyes; Drug: Vehicle to be administered in both eyes
- Treatment with Schirmer test with anesthetic (Experimental): Both eyes will be treated.
  Interventions: Drug: 0.003% AR-15512 to be administered in both eyes; Drug: Vehicle to be administered in both eyes

INTERVENTIONS:
Drug: 0.003% AR-15512 to be administered in both eyes — Two rounds of Schirmer tests, performed without anesthetic (per randomization), before and after instillation of 0.003% AR-15512
  Arms: Treatment with Schirmer test with no anesthetic
Drug: Vehicle to be administered in both eyes — Two rounds of Schirmer tests, performed without anesthetic, before and after instillation of Vehicle
  Arms: Treatment with Schirmer test with no anesthetic
Drug: 0.003% AR-15512 to be administered in both eyes — Two rounds of Schirmer tests, performed with anesthetic (per randomization), before and after instillation of 0.003% AR-15512
  Arms: Treatment with Schirmer test with anesthetic
Drug: Vehicle to be administered in both eyes — Two rounds of Schirmer tests, performed with anesthetic (per randomization), before and after instillation of Vehicle
  Arms: Treatment with Schirmer test with anesthetic

SUMMARY:
This will be a vehicle-controlled, masked, randomized study conducted at a single site in the United States. All participants enrolled will have Dry Eye Disease (DED). The study will consist of 2 Visits. At Visit 1, eligibility will be assessed at Screening. All eligible subjects will then be enrolled and randomized to one of two treatment groups (1:1): active (0.003% AR-15512) or control (AR-15512 vehicle). Subjects in each treatment group will then be randomized 1:1 to which Visit (Visit 1 or 2) anesthetic will be used with the Schirmer test.

ELIGIBILITY:
Inclusion Criteria:

* Have used, and/or desired to use artificial tears for DED symptoms within 6 months prior to Visit 1
* Within the last year from Visit 1, have a documented Schirmer test with or without topical anesthesia score ≥ 2 and ≤ 10 mm/5 min
* Within the last year from Visit 1, have documented symptoms of DED
* Corrected Visual Acuity (Snellen) 20/200 or better in both

Exclusion Criteria:

* Use of artificial tears within 2 hours prior to Visit 1
* Use of ocular cyclosporine or other prescription ophthalmic solution for DED (e.g., Restasis®, Cequa®, Xiidra®) within 30 days of Visit 1 or anticipated use during the study period.
* Regular use of any topical ocular non-DED medication or use of a topical ocular non-DED medication within 2 hours of Visit 1
* Use of contact lenses in either eye within 7 days prior to the Screening visit or planned use during the study
* Punctal or intracanalicular plug present in either eyelid or anticipated plug insertion or occlusion at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Unanesthetized Schirmer test | Day 1
  Proportion of subjects ≥ 10 mm increase in unanesthetized Schirmer score
  Schirmer strips placed, without anesthesia, in both eyes measure the amount of tear wetting over a 5 minute period, measured in whole millimeters to a maximum score of 35 mm. An ≥ 10 mm score indicates a better outcome.
Unanesthetized Schirmer test | Day 1
  Mean change in Unanesthetized Schirmer score
  Schirmer strips placed, without anesthesia, in both eyes measure the amount of tear wetting over a 5 minute period, measured in whole millimeters to a maximum score of 35 mm. A greater mean change indicates a better outcome.
Unanesthetized Schirmer test | Day 1
  Mean Unanesthetized Schirmer score
  Schirmer strips placed, without anesthesia, in both eyes measure the amount of tear wetting over 5 minute period, measured in whole millimeters to a maximum score of 35 mm. A greater mean value indicates a better outcome.
Anesthetized Schirmer test | Day 1
  Proportion of subjects ≥ 10 mm increase in anesthetized Schirmer score
  Schirmer strips placed with anesthesia, in both eyes measure the amount of tear wetting over a 5 minute period, measured in whole millimeters to a maximum score of 35 mm. An ≥ 10 mm score indicates a better outcome.
Anesthetized Schirmer test | Day 1
  Mean change in anesthetized Schirmer score.
  Schirmer strips placed without anesthesia, in both eyes measure the amount of tear wetting over a 5 minute period, measured in whole millimeters to a maximum score of 35 mm. A greater mean change indicates a better outcome.
Anesthetized Schirmer test | Day 1
  Mean anesthetized Schirmer score
  Schirmer strips placed with anesthesia, in both eyes measure the amount of tear wetting over 5 minute period, measured in whole millimeters to a maximum score of 35 mm. A greater mean value indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Senchyna, PhD, Study Director — Aerie Pharmaceuticals
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No